CLINICAL TRIAL: NCT06053047
Title: Remote Use of Thermovisual Monitoring to Reduce the RAte of Re-Ulceration in PatientS at Risk of RecurrenT Diabetic Foot UlcERs
Brief Title: Remote Monitoring of the Diabetic Foot to Prevent Re-Ulceration
Acronym: MASTER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsustainable recruitment rate - too slow to enroll participants
Sponsor: Bluedrop Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BMS CP002
Record Dates: First submitted 2023-09-12; First posted 2023-09-25 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot
Keywords: Diabetic Foot Ulcer (DFU); Remote monitoring; Telemedicine
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Use of Bluedrop Monitoring Service (Experimental): The BMS is made up of the Delta Foot Scanner (DFS) device, its accompanying Sentinel Review Interface (SRI) software and a Bluedrop virtual monitoring service.
  The DFS is intended to be used for 30 seconds, once per day, by a person in their home. It is important that while using the device that the participant continues with their routine foot care as recommended by their doctor.
  Interventions: Device: Bluedrop Monitoring Service (BMS)
- Standard of care (No Intervention): Participants continue with routine foot care as recommended by their doctor

INTERVENTIONS:
Device: Bluedrop Monitoring Service (BMS) — Remote use of ThermoVisual monitoring
  Arms: Use of Bluedrop Monitoring Service

SUMMARY:
The purpose of this study is to understand the effects of the Bluedrop Monitoring System (BMS) on the development of diabetic foot ulcers.

All Participants in this study will continue with their normal foot care and complete surveys with questions about their foot health every three months.

Participants selected to receive the Bluedrop Monitoring System (BMS) will place it in their home and stand on it once a day for 12 months. Participants will also need to answer questions about their general foot health and, if using the system, their experience using the device and monitoring service.

DETAILED DESCRIPTION:
This is a siteless study, which is planned to enroll approximately 200 patients with diabetes mellitus and a foot ulcer which has healed within 2-24 months prior to screening. The study will be organized and conducted via a central coordinating center at the Duke Clinical Research Institute. Potentially eligible patients within the state of North Carolina will be contacted about the study and if willing, will provide consent to participation remotely, including use of the Pluto Health''s unified medical records platform. Participants will not attend study sites, as all study visits will take place virtually and/or by telephone contact from the coordinating center and the primary study outcomes will be ascertained by review of health records via the Pluto system.

All enrolled participants will be randomized to use of the Bluedrop Monitoring System (BMS) or not in addition to their otherwise usual care. Participants assigned to use of the Bluedrop Monitoring System (BMS) will be provided the Delta Foot Scanner device with monitoring system and will be instructed in daily device use by Bluedrop personnel.

Participants will continue to receive all other usual care during the study period, and the patient's other care may be adjusted as considered clinically appropriate by the usual care provider(s).

After study enrollment, study visits will take place at 3, 6, 9 and 12 months. These visits will include participant surveys including assessment of neuropathy-specific quality of life, and review of health records via the Pluto Health platform by the study Principal Investigator (PI) to identify the occurrence of foot injury or ulcer and any associated medical or surgical care.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding of the study procedures and conditions of the protocol and agreement to participate in the study by providing consent prior to any study-specific procedures.
2. Male or female patients 18 years or older.
3. Diagnosis of type 1 or type 2 diabetes mellitus more than 3 months prior to the Screening Visit.
4. History of healed diabetic foot ulcer(s), present for at least 2 weeks and healed within 2-24 months prior to screening.
5. Confirmation of presence of peripheral neuropathy with loss of protective sensation (documented in medical records or certain ICD-10 codes for care of patients with diabetes and loss of protective sensation)
6. Patient has signed up for and provided or will provide consent to review of medical records available via the Pluto platform.
7. Access to internet service at the site of device use or willing to use a 4G router provided by the Sponsor
8. Access to cell phone on which they can receive study communications
9. Has a healthcare provider who is confirmed to be their point of contact for foot care or injuries and this HCP uses an EHR that is compatible with Pluto
10. English speaking

Exclusion Criteria:

1. Patients with active foot ulcers or other open foot lesions
2. Weight, when fully clothed, of greater than 150 kg
3. Active Charcot arthropathy defined as the phase where the foot is undergoing collapse
4. Active foot infection or gangrene
5. Any history of major or minor lower limb amputation of more than 3 toes. NOTE: the hallux toe must be present on both feet to be eligible
6. Critical limb ischemia as evidenced by rest pain. NOTE: a healed ulcer indicates adequate perfusion and qualifies for the study
7. End-stage kidney disease (estimated GFR <15 mL/min/1.73 m2, and/or receiving renal replacement therapy)
8. Known pregnancy at the time of enrollment.*
9. Any mental health disorder, psychiatric disorder, or alcohol or drug abuse history such that, in the opinion of the investigator, the patient is unreliable as a study participant
10. Any travel plans expected to result in an interruption of BMS use for greater than 30 consecutive days.
11. Unable to identify and/or return to a usual care provider for foot care for the duration of the study
12. Unable or unwilling to be enrolled in the Pluto unified medical records system
13. Other issue that, at the discretion of the PI, renders the participant ineligible for participation. This includes inability to use the BMS for at least 3 days per week.

    * Participants who become pregnant during the study will not be removed. Pregnancy will be noted in their mobile application profile and their participation in the study will be closely monitored.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Relative risk reduction in the incidence of new Diabetic Foot Ulcers (DFUs) | Up to 12 months
  Relative risk reduction in the incidence of new Diabetic Foot Ulcers (DFUs) (Wound Stage 2 or 3 as defined by University of Texas Staging System for Diabetic Foot Ulcers where a higher score is a worse outcome <min score of 0 and max score of 3>) in participants assigned to use of the BMS compared to those not assigned to use of the BMS

SECONDARY OUTCOMES:
Participant engagement rates in the Bluedrop Monitoring System (BMS) | Up to 12 months
  Defined as the percentage of participants whose average weekly adherence exceeds 3 days per week
Relative risk reduction in the severity of new Diabetic Foot Ulcers (DFUs) | Up to 12 months
  Relative risk reduction in the severity of new Diabetic Foot Ulcers (DFUs) in participants assigned to use of the BMS compared to those not assigned to use of the BMS
Relative risk reduction in resource utilization | Up to 12 months
  Both all-cause and related to diabetic foot complications, in participants assigned to use of the Bluedrop Monitoring System (BMS) compared to those not assigned to use of the Bluedrop Monitoring System (BMS)

OTHER OUTCOMES:
Improvement in participant-reported neuropathy-specific quality of life measures | Up to 12 months
  Survey-ascertained (improvement, better overall score) participant-reported neuropathy-specific quality of life measures
Healthcare Provider acceptance of Bluedrop Monitoring System (BMS) | Up to 12 months
  Survey-ascertained healthcare provider acceptance of Bluedrop Monitoring System (BMS) in the management of patients with prior Diabetic Foot Ulcer (DFU)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Green, MD, Principal Investigator — Duke UMC
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No